CLINICAL TRIAL: NCT03083418
Title: The Effect of External Diaphragmatic Pacemaker(EDP) on Diaphragmatic Function and Neural Respiratory Drive in Patient With Acute Exacerbation of Chronic Obstructive Pulmonary Disease(AECOPD)
Brief Title: The Effect of EDP on Diaphragmatic Function and Neural Respiratory Drive in Patient With AECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX20161020
Record Dates: First submitted 2016-12-27; First posted 2017-03-20 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2018-01

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Keywords: AECOPD; EDP; Neural Respiratory Drive; Surface EMGdi
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Experimental): No EDP treatment.
  Interventions: Device: control group
- EDP therapy group (Experimental): 30 minutes continuous stimulation each time, two times a day, a total of one weeks of treatment .Parameters: 30min stimulation time, pacing frequency of 9 beats / min, pulse frequency is 40 hertz, the stimulus intensity (output pulse amplitude) is in the range of 0~30 units, which should be adjusted according to the daily maximum tolerance (patients with no pain and tension).
  Interventions: Device: EDP

INTERVENTIONS:
Device: control group — No EDP treatment
  Arms: Control group
Device: EDP — Turn on the device, and clean the skin where the patch will be located according to the screen tip. Paste the two groups of small electrodes to the inferior 1/3 of the outer edge of bilateral sternocleidomastoid, and the large electrodes are pasted to the corresponding 2nd intercostal skin surface of pectoralis major at midclavicular line.Adjusting the stimulus intensity according to the daily maximum tolerance (patients with no pain and tension).30 minutes continuous stimulation each time, twice a day, a total of one weeks of treatment .
  Arms: EDP therapy group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common respiratory disease characterized by airflow limitation that is progressive and not fully reversible. Patients with acute exacerbation of COPD must be hospitalized, as for further increase in airway resistance, pulmonary alveolar excessive expansion, diaphragm fatigue and neural respiratory drive. In recent years, Pulmonary rehabilitation is recognized as a core component in the comprehensive management of COPD, EDP as a means of rehabilitation can alleviate diaphragmatic fatigue, improve ventilation function, reduce the neural respiratory drive in patients with COPD during hospitalization, but still lack of evidence based medicine. Surface EMGdi can accurately evaluate neural respiratory drive, its detection is non-invasive, simple and safety .Therefore,Neural respiratory drive by surface EMGdi can be used as an important index for evaluating the therapeutic efficacy of AECOPD patients during hospitalization.

In the present study, about 40 patients with COPD will be recruited as research subjects .And the investigators aim to explore the effect of EDP on diaphragmatic function and neural respiratory drive in patient with AECOPD.Contrast analysis will be conducted to evaluate the effects of EDP on patients with AECOPD, which may provide a reasonable basis for the clinical application of EDP to AECOPD patients.

DETAILED DESCRIPTION:
Patients with AECOPD will participate in a rehabilitation program for one week. Participants in the proposed study will be randomly divided into two intervention groups:controlgroup and EDP therapy group. Before using EDP,the investigators will measure the relevant parameters of lung volume , diaphragm electromyogram, diaphragm activity and other basline index. Then EDP will be applied to investigate the effects of EDP on the above mentioned respiratory mechanics parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary function test of forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70% after inhalation of bronchial dilation agent.
* Patients in a clinically acute exacebation state.

Exclusion Criteria:

* Patients were excluded if they had evidence of pneumothorax or mediastinal emphysema and pacemaker installed.
* Patients with acute cardiovascular event and severe cor pulmonale.
* Patients with poor compliance.
* An Other causes of diaphragmatic dysfunction.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function(composite outcome measure) | Change from baseline in diaphragm electromyogram.(1 week later)
  Diaphragmatic function can be assessed by surface diaphragm electromyogram (EMGdi), which reflect the physiological activity of the diaphragm and indicate functional status of the neural respiratory drive.

SECONDARY OUTCOMES:
Degree of dyspnea(composite outcome measure) | Change from baseline in degree of dyspnea.(1 week later)
  Difference in the degree of dyspnea can be measured by borg index.
Pulmonary Function(composite outcome measure) | Change from baseline in pulmonary function.(1 week later)
  Pulmonary function is measured using a spirometer(PonyFX 229, Cosmed, Rome, Italy) that is calibrated daily.The FEV1 and percent-of-predicted FEV1, FVC and percent-of-predicted FVC which are presented in one report are used to evaluate Pulmonary Function.
Exercise Capacity(composite outcome measure) | Change from baseline in exercise capacity.(1 week later)
  Exercise capacity is evaluated using the 6-min walking distance (6MWD) according to American Thoracic Society guidelines.
Diaphragm activity(composite outcome measure) | Change from baseline in diaphragm activity.(1 week later)
  The degree of activity of the left and right diaphragmatic muscles in the general breath and deep breath were measured respectively.
Diaphragm thickness(composite outcome measure) | Change from baseline in diaphragm thickness.(1 week later)
  The changes of diaphragm thickness of the left and right diaphragmatic muscles in the breath were measured respectively.
Inspiratory muscle function(composite outcome measure) | Change from baseline in inspiratory muscle function.(1 week later)
  Currently, the maximal inspiratory pressure (PImax) and maximal expiratory pressures(PEmax) are measured by a digital manometer (AZ-8205, AZ Instrument, Taichung City, Taiwan)and combined to evaluate inspiratory muscle function.

OTHER OUTCOMES:
Body Composition Monitor(composite outcome measure) | Change from baseline in body composition.(1 week later)
  Body composition abnormalities are prevalent in COPD.Human body composition analyzer can detect various elements of human body and analyze human health status.
Health-related quality(composite outcome measure) | Change from baseline in health-related quality.(1 week later)
  Health-related quality is a component of the broader concept of quality of life and is defined as satisfaction with health.The St. George's Respiratory Questionnaire (SGRQ) and Chronic Respiratory Disease Questionnaire (CRQ）;and its self-reported version are the most widely used disease-specific questionnaires.
Symptom Evaluation(composite outcome measure) | Change from baseline in symptom evaluation.(1 week later)
  Individuals with chronic respiratory disease often have symptoms such as dyspnea, fatigue, cough, weakness,sleeplessness,and psychological distress.Instruments for assessment of multiple symptoms include COPD Assessment Test (CAT) and Modified Medical British Research Council Scale(mMRC).

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No